CLINICAL TRIAL: NCT02180698
Title: A Phase I Study to Determine the Safety of the Combination of Stable-Emulsion Formulation of Glucopyranosyl Lipid A (GLA-SE) With Radiation in Patients With Metastatic Sarcoma
Brief Title: TLR4 Agonist GLA-SE and Radiation Therapy in Treating Patients With Soft Tissue Sarcoma That Is Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9145; NCI-2014-01299 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9145 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy; Radiation; glucopyranosyl lipid-A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (TLR4 agonist GLA-SE, radiation therapy) (Experimental): Patients receive TLR4 agonist GLA-SE intratumorally once weekly for 8 weeks. Within 2 weeks of starting treatment, patients also undergo radiation therapy over 2 weeks for a total of 5-6 fractions.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy; Drug: TLR4 Agonist GLA-SE

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: TLR4 Agonist GLA-SE — Given intratumorally
  Other Names: GLA-SE; Glucopyranosyl Lipid A in Stable Emulsion; Glucopyranosyl Lipid Adjuvant-Stable Emulsion; Toll-like Receptor 4 Agonist GLA-SE

SUMMARY:
This pilot phase I clinical trial studies the side effects and best dose of toll-like receptor 4 (TLR4) agonist glucopyranosyl lipid A (GLA)-stable-emulsion (SE) when given together with radiation therapy in treating patients with soft tissue sarcoma that has spread to other parts of the body (metastatic) or cannot be removed by surgery (unresectable). TLR4 agonist GLA-SE may stimulate the immune system to kill sarcoma cells. Radiation therapy uses high energy x rays to kill tumor cells. Giving TLR4 agonist GLA-SE with radiation therapy may be a better treatment to treat sarcoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of weekly injections of GLA-SE (TLR4 agonist GLA-SE) in combination with palliative radiation in patients with metastatic sarcoma.

SECONDARY OBJECTIVES:

I. To look for preliminary evidence of efficacy at distant tumor sites following the combination of radiation and intra-tumor injection of GLA-SE.

II. To analyze changes in tumor-immune infiltrates following radiation and intra-tumor injection of GLA-SE.

OUTLINE: This is a dose-escalation study of TLR4 agonist GLA-SE.

Patients receive TLR4 agonist GLA-SE intratumorally once weekly for 8 weeks. Within 2 weeks of starting treatment, patients also undergo radiation therapy over 2 weeks for a total of 5-6 fractions.

After completion of study treatment, patients are followed up every 6 weeks for 6 months and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of metastatic or unresectable sarcoma
* Patient must have a palpable, superficial tumor, safely accessible for bedside injection that will be radiated and can be accurately localized and stabilized if needed
* Patient must have consulted with a radiation oncologist who is planning radiation; radiation should be completed within a 2-week window from start to finish
* Patient must be willing to undergo biopsies as specified by the protocol; the biopsy requirement can only be waived if deemed unsafe by the patient's treating physician or the principal investigator (PI)
* Zubrod (Eastern Cooperative Oncology Group [ECOG]) performance status of '0-2'
* Serum creatinine =< 1.5 times the upper limit of normal
* Total bilirubin =< 1.5 times the upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times the upper limit of normal
* Prothrombin time (PT) =< 1.5 times the upper limit of normal
* Partial thromboplastin time (PTT) =< 1.5 times the upper limit of normal
* Absolute neutrophil > 1000/uL
* Platelet count > 75,000/uL
* For patients who will be entering the "expansion phase" of the trial, the patient must be able to safely delay radiation by at least 6 weeks

Exclusion Criteria:

* Pregnant women, nursing women, men and women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to study entry
* Known active symptomatic congestive heart failure
* Known clinically significant hypotension
* Known newly diagnosed cardiac arrhythmia; patients with an arrhythmia that has been stable for at least 3 months will be allowed to participate
* Known untreated central nervous system (CNS) metastasis
* Patients with known systemic infections requiring antibiotics or chronic maintenance/suppressive therapy
* Systemic anticancer therapy (chemotherapy, "biologics", immunotherapy) less than two weeks prior to starting radiation
* Known clinically significant autoimmune disorders requiring on-going systemic immune-suppression for control
* Current treatment with steroids
* Patients who are known to be human immunodeficiency virus (HIV) positive must have a normal cluster of differentiation (CD)4 count and undetectable viral load
* Current treatment with warfarin; for patients not on an anti-platelet agent such as aspirin, other anticoagulation is acceptable so long as the treating physician feels that it is safe to hold it on the day of the biopsy until after the biopsy has been safely completed
* Known allergy(ies) to any component of the study agent GLA-SE including egg lecithin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

PRIMARY OUTCOMES:
Incidence of severe adverse events, defined as any grade 3 or higher adverse event (AE) according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to week 9
  The highest toxicity grades per patient will be tabulated for AEs and laboratory measurements as will the numbers and percentages of patients reporting AEs.

SECONDARY OUTCOMES:
Change in biomarker outcomes from the peripheral blood | Baseline up to 1 year
  Summary statistics will be used to describe changes across time. In addition, the time course of biomarker outcomes from the peripheral blood will be investigated graphically, by summary plots or individual patient plots. If there is suggestion of meaningful trend, methods such as linear mixed models may be used to characterize the pattern of change over time.
Clinical benefit based on RECIST v1.1 and iRRC evaluations | Up to 1 year
  Categorical data analysis and logistic regression will be used to evaluate the associations between correlative measures and clinical outcome (e.g., response, clinical benefit, time to progression, progression-free survival, and survival).
Immune infiltrates, measured quantitatively as number of cells per unit area | Up to 1 year
  Tumor infiltrating lymphocytes will be analyzed directly by flow and grown in vitro so that functional characteristics can be analyzed. Metrics based on flow cytometry (e.g. cell phenotype and inhibitory receptor expression) will be reported both with respect to the mean florescence intensity of the staining as well as the absolute and relative numbers of positive and negative cells compared with established controls.
Progression free survival | Up to 1 year
  Categorical data analysis and logistic regression will be used to evaluate the associations between correlative measures and clinical outcome (e.g., response, clinical benefit, time to progression, progression-free survival, and survival). Kaplan-Meier methodology and Cox Proportional Hazards models will be used to evaluate time-to-event endpoints.
Response based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 and immune-related-response criteria (iRRC) evaluations | Up to 1 year
  Categorical data analysis and logistic regression will be used to evaluate the associations between correlative measures and clinical outcome (e.g., response, clinical benefit, time to progression, progression-free survival, and survival).
Survival | Up to 1 year
  Categorical data analysis and logistic regression will be used to evaluate the associations between correlative measures and clinical outcome (e.g., response, clinical benefit, time to progression, progression-free survival, and survival). Kaplan-Meier methodology and Cox Proportional Hazards models will be used to evaluate time-to-event endpoints.
Time to progression | Up to 1 year
  Categorical data analysis and logistic regression will be used to evaluate the associations between correlative measures and clinical outcome (e.g., response, clinical benefit, time to progression, progression-free survival, and survival). Kaplan-Meier methodology and Cox Proportional Hazards models will be used to evaluate time-to-event endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pollack, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Seo YD, Lu H, Black G, Smythe K, Yu Y, Hsu C, Ng J, Hermida de Viveiros P, Warren EH, Schroeder BA, O'Malley RB, Cranmer LD, Loggers ET, Wagner MJ, Bonham L, Pillarisetty VG, Kane G, Berglund P, Hsu FJ, Mi X, Alexiev BA, Pierce RH, Riddell SR, Jones RL, Ter Meulen J, Kim EY, Pollack SM. Toll-Like Receptor 4 Agonist Injection With Concurrent Radiotherapy in Patients With Metastatic Soft Tissue Sarcoma: A Phase 1 Nonrandomized Controlled Trial. JAMA Oncol. 2023 Dec 1;9(12):1660-1668. doi: 10.1001/jamaoncol.2023.4015. PMID 37824131
- [Derived] Goff PH, Riolobos L, LaFleur BJ, Spraker MB, Seo YD, Smythe KS, Campbell JS, Pierce RH, Zhang Y, He Q, Kim EY, Schaub SK, Kane GM, Mantilla JG, Chen EY, Ricciotti R, Thompson MJ, Cranmer LD, Wagner MJ, Loggers ET, Jones RL, Murphy E, Blumenschein WM, McClanahan TK, Earls J, Flanagan KC, LaFranzo NA, Kim TS, Pollack SM. Neoadjuvant Therapy Induces a Potent Immune Response to Sarcoma, Dominated by Myeloid and B Cells. Clin Cancer Res. 2022 Apr 14;28(8):1701-1711. doi: 10.1158/1078-0432.CCR-21-4239. PMID 35115306